CLINICAL TRIAL: NCT05946551
Title: Feasibility Assessment of a Decentralized Platform Adaptive Double-Blind, Randomized Controlled Trial Investigating Repurposed Drugs in the Treatment of Post-Acute Sequelae of Coronavirus-19 (PASC)
Brief Title: Treatment of Long CoronaVirus Disease (COVID) (TLC) Feasibility Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to lack of funding.
Sponsor: Emory University (Other)
Collaborators: CURE Drug Repurposing Collaboratory (CDRC) (Unknown)
Responsible Party: Principal Investigator, Tiffany A Walker, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00005537
Record Dates: First submitted 2023-07-12; First posted 2023-07-14 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: Long COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Cetirizine; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HRA Treatment Arm (Experimental): Participants randomized to Treatment Arm will receive dual histamine receptor antagonists: famotidine and cetirizine daily.
  Interventions: Drug: Cetirizine; Drug: Famotidine
- Placebo Arm (Placebo Comparator): The compounding study pharmacy will provide placebo capsules to the patients randomized to Placebo. These capsules are manufactured to match each treatment drug for oral administration.
  Interventions: Drug: Cetirizine Placebo; Drug: Famotidine Placebo

INTERVENTIONS:
Drug: Cetirizine — Cetirizine will be dispensed as a 10mg capsule with instructions for patients to take one capsule daily by mouth, preferably at bedtime.
  Arms: HRA Treatment Arm
Drug: Famotidine — Famotidine will be dispensed in 20mg capsules with instructions for patients to take one capsule twice daily, as close to the same times every day as possible.
  Other Names: HRA
  Arms: HRA Treatment Arm
Drug: Cetirizine Placebo — The cetirizine placebo will be designed as a capsule of an inert substance and will match the morphology of the cetirizine treatment capsule. Administration instructions to match that of cetirizine.
  Arms: Placebo Arm
Drug: Famotidine Placebo — The famotidine placebo will be designed as a capsule of an inert substance and will match the morphology of the famotidine treatment capsule. Administration instructions to match that of famotidine.
  Arms: Placebo Arm

SUMMARY:
The primary objective of this study is to assess the feasibility and acceptability of methods and procedures to be employed in a larger scale decentralized platform adaptive randomized clinical trial in patients with a history of a Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Polymerase Chain Reaction (PCR) positive test and/or medical records from a healthcare provider that coincides with the diagnosis of long-COVID.

DETAILED DESCRIPTION:
Fully decentralized single-center, double-blind, randomized, placebo-controlled pilot feasibility trial for patients reporting symptoms consistent with at least one of the following PASC symptoms: Brain fog, Fatigue, Headache, Sleep Disturbance, Post-exertional Malaise (PEM), or Dysautonomia.

Participants' interactions with study staff and the study visits will occur primarily via REDCap and Zoom. Informed consent will be conducted remotely via Zoom and obtained electronically in REDCap. Subjects will complete protocol-required logs, questionnaires, and surveys in REDCap. Dose tolerability assessments will occur via televisit preferably, or phone if necessary.

Following informed consent, subjects will enter a 4-week screening period during which medical records will be obtained and reviewed. At baseline (Day -28) subjects will complete a battery of tests consisting of the World Health Organization Disability Assessment Schedule (WHODAS) 2.0, Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue 7a, Insomnia Severity Scale, PROMIS Cognitive Function 6A, DePaul Symptom Questionnaire - Post-Exertional Malaise (DSQ-PEM) Short Form, Headache Diary, COMPASS 31, and Self-reported persistent symptoms questionnaire. The headache diary requires daily tracking for 7 days (i.e., Day -28- Day -22).

Subjects who complete the screening phase will proceed to randomization where they will be randomized 2:1 to either histamine receptor antagonists (cetirizine and famotidine) or matching placebos. Emory University's Investigational Drug Services (IDS) will conduct the randomization and will overnight via national courier the assigned medication to the study subject. The treatment phase of 12 weeks starts upon ingestion of the first dose.

Cetirizine and famotidine will be supplied as 10mg capsules and 20mg capsules respectively. Dosing for the entire treatment period is one 10mg capsule cetirizine or placebo once daily, preferably at bedtime, and one 20mg capsule famotidine or placebo twice daily, as near as possible to the same time every day. Dose tolerability will be assessed on Day 14 via televisit or phone call. If the dose of either IP is not tolerated, subjects will be removed from the study. If the doses are tolerated, subjects will be resupplied and tolerability assessed per protocol.

Throughout the treatment phase subjects in all arms will complete the symptom questionnaire, adverse event, study drug adherence, and concomitant medication logs weekly. All subjects will complete the full battery of tests on Days 42, 63, and 84 (Weeks 6, 9, and 12). Subjects will have a +/- 3-day window in which to complete the battery. However, the headache diary requires daily tracking for the 7 days preceding Days 43, 63, and 84. On Day 84 all subjects will complete an end-of-study survey assessing their thoughts and feelings about the study methods and procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age with a history of a SARS-CoV-2 PCR positive test and/or medical records from a healthcare provider that coincides with the diagnosis of long-COVID
2. New or worsened symptoms since the onset of COVID-19 that are persistent at the time of enrollment and have lasted for ≥ 12 weeks (including at least one of the following: fatigue, post-exertional malaise (PEM), headache, brain fog, sleep disturbance, dysautonomia.
3. Confirmation of negative urine or serum human chorionic gonadotropin (HCG) (pregnancy) test in women of childbearing potential
4. Willing to use appropriate contraceptives for female and male subjects for the duration of the study
5. Has an address (for mailing of study drug) in the state of Georgia
6. Able to swallow capsules
7. Has reliable access to a mobile phone, tablet, laptop, or desktop computer capable of connecting to the internet via Wi-Fi or a data plan
8. Available lab work (CBC and CMP) after the onset of long COVID symptoms
9. Willing and able to comply with scheduled visits, treatment plan, and other study procedures including receiving either intervention or placebo
10. Willing to not take any of the study medications while enrolled in the study except for essential needs as prescribed by a healthcare provider

Exclusion Criteria:

1. No post-acute COVID-19 symptoms (PASC) symptoms at the time of enrollment or PASC symptoms present <12 weeks at the time of enrollment
2. Inability to provide own informed consent
3. Currently Hospitalized
4. For women of childbearing potential (WOCBP), currently pregnant or plans to become pregnant during the study period; for males with partners of childbearing potential (OCBP), plans to become pregnant during the study period
5. Actively enrolled in another Long COVID/PASC interventional trial or participation in another interventional clinical trial in the last 30 days or planned during the trial period
6. Unstable medical comorbidities (e.g., decompensated cirrhosis, stage III-IV chronic kidney disease, New York Heart Association (NYHA) class III congestive heart failure), per the patient report, telemedicine physical exam, baseline laboratory values (hematology and extended chemistry panels) and/or medical records
7. Other medical conditions occurring after the onset of COVID-19 that can otherwise account for PASC-type symptoms
8. Currently immunocompromised from the following: solid organ transplant, bone marrow transplant (BMT), high dose steroids (>20mg prednisone per day), immune modulators, or chemotherapy
9. Currently taking opioid analgesics, undergoing treatment for opioid addiction, or taking any other prohibited concomitant medication
10. Opioid dependence or withdrawal syndrome
11. Known sensitivity or adverse reaction to H1 or H2 receptor antagonists, or medication components
12. Suspected or confirmed pregnancy or breastfeeding
13. Participants already on H1 or H2 receptor antagonists within three (3) months of randomization
14. Currently receiving other therapies to treat COVID-19 or Long COVID symptoms, e.g., convalescent plasma, remdesivir, Paxlovid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Walker, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia
  - Metro-Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets may be available to external researchers following final analyses. Requests will be evaluated on a case-by-case basis by PI. No data will be released without proof of Institutional Review Board (IRB) approval or determination. Agreements as required by local policies will be completed when necessary.
Supporting Information: Study Protocol
Time Frame: Datasets may be available following final analyses and publication.
Access Criteria: Proposals should be directed to tiffany.austin.walker@emory.edu.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants were recruited from Emory and Grady Healthcare System in Atlanta, Georgia, USA. Participant enrollment began on March 08, 2024, and follow-up for the five participants was complete by June 24, 2024. The study was terminated due to a lack of funding.
Period: Overall Study
Arm/Group | HRA Treatment Arm | Placebo Arm
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRA Treatment Arm | Placebo Arm | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had Any Confusion Over How to Take the Study Drug, Including Which Pill to Take, When to Take it, or How Many to Take
Description: The number of participants that had any confusion over how to take the study drug, including which pill to take, when to take it, or how many to take will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

2. Primary Outcome: Number of Participants That Had Trouble Adhering to the Study Drug Schedule
Description: The number of participants that had trouble adhering to the study drug schedule will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

3. Primary Outcome: Number of Participants That Had Any Difficulty Using the REDCap Interface.
Description: The number of participants that had any difficulty using the REDCap interface will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

4. Primary Outcome: Number of Participants That Prefer Participating in This Virtual Study
Description: The number of participants that prefer participating in this virtual study compared to participating in an in-person study hosted at a medical center will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

5. Primary Outcome: Number of Participants Satisfied With Their Opportunities to Interact With Study Staff
Description: The number of participants satisfied with their opportunities to interact with study staff will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

6. Primary Outcome: Number of Participants That Felt They Could Reach Study Staff if Needed
Description: The number of participants that felt they could reach study staff if needed will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

7. Primary Outcome: Number of Participants That Felt That Study Staff Was Available and Easy to Contact to Report Any Adverse Effects
Description: The number of participants that felt that study staff was available and easy to contact to report any adverse effects that they experienced from the medication will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

8. Primary Outcome: Number of Participants That Felt That the Amount of Information Collected in Each Series of Surveys Was Acceptable
Description: The number of participants that felt that the amount of information collected in each series of surveys was acceptable will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

9. Primary Outcome: Number of Participants That Felt That the Frequency in Which the Information Was Collected Was Acceptable
Description: The number of participants that felt that the frequency in which the information was collected was acceptable will be recorded as part of the end-of-study survey.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

10. Primary Outcome: Improvement Rating
Description: Participants will be asked how much they feel they improved from this treatment over the last 12 week using a scale from 1 to 5, with 5 being complete improvement (better outcome) and 1 being no improvement.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Score on a scale | 2.3 (0.94) | 2 (0)

11. Primary Outcome: Quality of Life (QoL) Score Rating
Description: Participants will be asked how much their quality of life was impacted by changes to their health during the study. On a scale of 1 to 5 with 5 being the most impacted (better outcome) and 1 being not at all impacted by changes to their health.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Score on a scale | 2 (1.4) | 1.5 (0.5)

12. Primary Outcome: Interest Score
Description: Participants will be asked how interested they are in continuing treatment with the study medication after the study. On a scale of 1 to 5, with 5 being completely interested (better outcome) and 1 being completely uninterested.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
score on a scale | 4.3 (0.94) | 3 (2)

13. Secondary Outcome: Proportion of Survey Completion
Description: Percentage of participants who complete 70% of surveys will be assessed
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

14. Secondary Outcome: Proportion of Study Drug Adherence
Description: Percentage of participants who complete 70% of doses will be assessed
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

15. Secondary Outcome: Proportion of Lost to Follow Up (LFUP)
Description: Percentage of participants Lost to Follow Up (LFUP) will be assessed
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

16. Secondary Outcome: Proportion of Voluntary Termination
Description: Percentage of participants that voluntarily terminate participation will be assessed
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

17. Secondary Outcome: Adverse Events (AEs) Incidence
Description: The mean number of adverse events in the treatment arms will be compared to those in the placebo arm.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Mean (Standard Deviation); unit: number of adverse events
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
number of adverse events | 3.7 (1.2) | 2 (1)

18. Secondary Outcome: Serious, Unexpected Suspected Adverse Reactions (SUSAR) Incidence
Description: The number of SUSARs in the treatment arms versus the placebo arm will be recorded.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Number; unit: Number of SUSARs
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Number of SUSARs | 0 | 0

19. Secondary Outcome: Study-wide Serious Adverse Events (SAEs) Incidence
Description: The total number of SAEs in the treatment arms versus the placebo arm will be recorded.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Number; unit: Number of SAEs
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Number of SAEs | 0 | 0

20. Secondary Outcome: Number of Discontinuations or Temporary Suspensions of IP
Description: The total number of participants who discontinue any of the treatment arms versus the placebo arm will be recorded.
Time Frame: End of the Treatment Phase at 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HRA Treatment Arm | Placebo Arm
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events, Serious Adverse Effects were assessed after randomization until completion of the study (12 weeks post-intervention).
Arm/Group | HRA Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HRA Treatment Arm (N=3) | Placebo Arm (N=2)
Sore neck (Musculoskeletal and connective tissue disorders) | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Herpes Zoster (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT05946551/Prot_SAP_000.pdf